CLINICAL TRIAL: NCT02713659
Title: Early Literacy Promotion Among Poor Urban Children in Philadelphia
Brief Title: Early Literacy Promotion Intervention
Acronym: ELPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: William Penn Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 15-012507
Record Dates: First submitted 2016-03-10; First posted 2016-03-21 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Child Development
Keywords: Literacy; Child Development; Reading
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Literacy Promotion (Experimental): Parents and children randomized to the Early Literacy Promotion arm.
  Interventions: Behavioral: Early Literacy Promotion
- Standard Literacy Promotion (Active Comparator): Parents and children randomized to the Standard Literacy Promotion arm.
  Interventions: Behavioral: Standard Literacy Promotion

INTERVENTIONS:
Behavioral: Early Literacy Promotion — Parents will receive a book with developmentally appropriate advice about reading at each well child visit from one week through 5 months of age, as well as weekly text reminders related to reading. From 6 months of age, both groups will receive standard literacy promotion and will attend study visits every six months until age 2.
  Arms: Early Literacy Promotion
Behavioral: Standard Literacy Promotion — Parents will receive weekly text messages about child safety, and no books before the age of 6 months from their provider. From 6 months of age, both groups will receive standard literacy promotion and will attend study visits every six months until age 2.
  Arms: Standard Literacy Promotion

SUMMARY:
This study is testing the effects of early literacy promotion compared to standard literacy promotion at The Children's Hospital of Philadelphia. Eligible participants and their families will be consented and randomly assigned into either a standard literacy program or an early literacy program. Standard literacy will consist of the receipt of books and reading promotion beginning at 6 months of age, while early literacy will consist of the receipt of books and reading promotion beginning in the newborn period. In both groups, participants will receive weekly text messages until the child is 6 months old (the text messages will either about reading or safety) and have follow-up study visits at 6, 12, 18, and 24 months. The study will examine the effects of the intervention on language development and reading behaviors.

DETAILED DESCRIPTION:
Poor urban children are at an increased risk for language and cognitive delays. Such delays can lead to poor school readiness and disparities in educational outcomes when compared to children from middle and upper income strata. Reach Out and Read (ROR), a national program which promotes parent-child reading activities for children 6 months through 5 years of age at pediatric well child visits, has been shown to improve at-risk children's expressive and receptive language development. However, poor children who participate in ROR still demonstrate language outcomes that are below national averages. It isn't clear whether early literacy promotion, i.e. promotion of parent-child reading prior to six months of age, is more effective than standard literacy promotion and can further improve poor children's language and cognitive outcomes. Therefore, this study will test the effectiveness of early literacy promotion compared to standard literacy promotion among poor at-risk children. Children with Medicaid insurance who are under 1 month of age, were born at least 35 weeks gestation, whose mothers speak English or Spanish and are 15 years of age and older, and are without any neurodevelopmental disabilities will be eligible to participate. One to two urban practices affiliated with The Children's Hospital of Philadelphia (CHOP) who have implemented ROR as standard practice will be recruited to participate. One hundred twenty eligible children attending participating practices will be recruited to participate and consented, stratified by practice site, and randomized to receive early literacy promotion or standard literacy promotion. Early literacy promotion will consist of the provision of developmentally appropriate books selected specifically for well visits starting from one month of age to six months; discussion of the importance of reading, talking, and singing by pediatric clinicians; and text message reminders to parents concerning early literacy and daily reading. Standard literacy promotion will consist of the Reach Out and Read Program with provision of developmentally appropriate books at all well visits from six months of age onward and promotion of reading, talking, and singing activities by pediatric clinicians. Mothers will complete study measures consisting of demographic characteristics, postpartum depression symptoms, health literacy, and adverse childhood experiences at enrollment, and mothers and children will complete measures of reading activity (Stim-Q) at 6, 12, 18, and 24 months of age and child expressive and receptive language development (Preschool Language Scale) at 6 and 24 months of age. Differences in child language outcomes will be assessed using intention-to-treat. Results of this study will be disseminated to key stakeholders through peer-reviewed manuscripts, reports, social media, and evidence-to-action briefs prepared by Policylab at the Children's Hospital of Philadelphia. Study findings will be of importance to the Annie E. Casey Foundation's Read! By 4th in Philadelphia and other community Grade-Level Reading Campaigns, the Clinton Foundation's Too Small to Fail initiative to advance early brain development, and Great Start Collaborative's Early to Read campaign.

ELIGIBILITY:
Inclusion Criteria:

1. English or Spanish speaking
2. Mothers 15 years of age or older at the start of the study
3. Child born ≥ 35 weeks estimated gestational age (EGA)
4. Child less than 4 weeks old at enrollment
5. Child with Medicaid Insurance

Exclusion Criteria:

1. Child born premature < 35 weeks EGA
2. Children with neurodevelopmental disabilities or congenital malformation at increased risk of language delays

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P Guevara, MD, MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Following completion of all analyses, data will be de-identified and made available for other investigators.
Supporting Information: Study Protocol
Time Frame: 12 months after publication of all relevant papers
Access Criteria: De-identified only

REFERENCES:
- [Derived] Guevara JP, Erkoboni D, Gerdes M, Winston S, Sands D, Rogers K, Haecker T, Jimenez ME, Mendelsohn AL. Effects of Early Literacy Promotion on Child Language Development and Home Reading Environment: A Randomized Controlled Trial. J Pediatr X. 2020 May 11;2:100020. doi: 10.1016/j.ympdx.2020.100020. eCollection 2020 Spring. PMID 37332625

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Literacy Promotion: Parents will receive a book with developmentally appropriate advice about reading at each well child visit from one week through 5 months of age, as well as weekly text reminders related to reading. From 6 months of age, this group will receive standard literacy promotion and will attend study visits every six months until age 2.
- Standard Literacy Promotion: Parents will receive weekly text messages about child safety, and no books before the age of 6 months from their provider. From 6 months of age, this group will receive standard literacy promotion and will attend study visits every six months until age 2.
Period: Baseline
Arm/Group | Early Literacy Promotion | Standard Literacy Promotion
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0
Period: 6 Month Study Visit
Arm/Group | Early Literacy Promotion | Standard Literacy Promotion
Started | 60 | 60
Completed | 53 | 47
Not Completed | 7 | 13
Period: 12 Month Study Visit
Arm/Group | Early Literacy Promotion | Standard Literacy Promotion
Started | 57 | 55
Completed | 54 | 52
Not Completed | 3 | 3
Period: 18 Month Study Visit
Arm/Group | Early Literacy Promotion | Standard Literacy Promotion
Started | 58 | 53
Completed | 50 | 50
Not Completed | 8 | 3
Period: 24 Month Study Visit
Arm/Group | Early Literacy Promotion | Standard Literacy Promotion
Started | 57 | 52
Completed | 49 | 44
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Literacy Promotion | Standard Literacy Promotion | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Enrollment Population: Numbers in columns may not sum to overall totals due to missing data.
  years
    Mother's Age | 25.4 (5.2) | 25.3 (5.2) | 25.4 (5.2)
    Father's Age: number analyzed (Participants) | 59 | 57 | 116
    Father's Age | 28.2 (6.4) | 28.7 (7.0) | 28.4 (6.7)
Age, Continuous [Mean (Standard Deviation); unit: Infant Age (Days)] — Infant Age in Days
  Infant Age (Days) | 5.4 (2.1) | 5.6 (2.3) | 5.5 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Child Gender: Female | 32 | 34 | 66
  Child Gender: Male | 28 | 26 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 57 | 46 | 103
  Race: White | 0 | 2 | 2
  Race: Hispanic | 2 | 4 | 6
  Race: Other | 1 | 8 | 9
Marital Status [Count of Participants; unit: Participants] — Population: Numbers in columns may not sum to overall totals due to missing data.
  Participants
    number analyzed (Participants) | 59 | 59 | 118
    Single | 40 | 39 | 79
    Married/Living Together as if Married | 17 | 20 | 37
    Seperated/Divorced | 2 | 0 | 2
Annual Household Income [Count of Participants; unit: Participants] — Population: Numbers in columns may not sum to overall totals due to missing data.
  Participants
    number analyzed (Participants) | 58 | 59 | 117
    $0 - $24,000 | 47 | 48 | 95
    $25,000 - $49,000 | 11 | 11 | 22
Education Level [Count of Participants; unit: Participants] — Population: Numbers in columns may not sum to overall totals due to missing data.
  Participants
    number analyzed (Participants) | 59 | 59 | 118
    Some High School | 11 | 9 | 20
    High School/GED | 27 | 24 | 51
    Some College | 18 | 23 | 41
    College/Post College Degree | 3 | 3 | 6
Number of Other Adults in the Household [Mean (Standard Deviation); unit: people] — Population: Numbers in columns may not sum to overall totals due to missing data.
  people
    number analyzed (Participants) | 60 | 59 | 119
    (all) | 1.3 (1.1) | 1.2 (0.6) | 1.3 (0.9)
Number of Other Children in the Household [Mean (Standard Deviation); unit: children] — Population: Numbers in columns may not sum to overall totals due to missing data.
  children
    number analyzed (Participants) | 60 | 59 | 119
    (all) | 1.2 (1.2) | 1.0 (1.2) | 1.1 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Preschool Language Scale-5th Edition Score
Description: The Preschool Language Scale-5th Edition (PLS) is a validated measure of expressive and receptive language function among children from birth through 7 years of age and is available in Spanish and English. PLS-5 provides three norm-referenced standard scores: Auditory Comprehension (AC) standard score, Expressive Communication (EC) standard score, and Total Language (TL) composite score. The scores are on a normalized standard score scale that has a mean of 100 and a standard deviation of 15 with scores ranging from 0-200. Higher scores represent better language development..
Time Frame: Change in PLS scores from 6 to 24 months of age
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Literacy Promotion | Standard Literacy Promotion
Number analyzed (Participants) | 49 | 44
score on a scale
  Difference in Auditory Standard Score | -8.2 (18.4) | -9.0 (16.5)
  Difference in Expressive Standard Score | -3.9 (15.6) | -2.0 (10.5)
  Difference in Total Standard Score | -5.9 (16.3) | -3.3 (19.0)
Statistical Analysis 1: Comparison: Early Literacy Promotion vs Standard Literacy Promotion; Auditory standard score between infants at 6 months and 24 months of age in the Early literacy arm and the standard literacy arm; Test type: Equivalence — 0.05; p = 0.85, t-test, 2 sided
Statistical Analysis 2: Comparison: Early Literacy Promotion vs Standard Literacy Promotion; Expressive standard score between infants at 6 months and 24 months of age in the Early literacy arm and the standard literacy arm; Test type: Equivalence — 0.05; p = 0.53, t-test, 2 sided
Statistical Analysis 3: Comparison: Early Literacy Promotion vs Standard Literacy Promotion; Total standard score between infants at 6 months and 24 months of age in the Early literacy arm and the standard literacy arm; Test type: Equivalence — 0.05; p = 0.49, t-test, 2 sided

2. Secondary Outcome: Change in StimQ Score
Description: Reading activity is measured using the StimQ Read Subscale, a subscale scale of the overall StimQ that measures the home reading environment among young children ages 5 to 36 months, and is available in Spanish and English. The Read Subscale of the StimQ-I is used for infants 5-12 months old and contains 12 questions, while the Read Subscale of the StimQ-T is used for children aged 12-36 months old and contains 11 questions. Scores range from 0-19 with higher scores representing better home reading environments.
Time Frame: Change in StimQ score from 6 to 24 months of age
Population: One participant only completed the StimQ survey at 24 months, therefore this number includes that participant. However, they are not counted in the total number of participants who completed the 24-month study visit because they did not complete the rest of the study visit surveys.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Early Literacy Promotion | Standard Literacy Promotion
Number analyzed (Participants) | 49 | 45
Scores on a Scale | 2.4 (3.2) | 2.8 (4.0)
Statistical Analysis 1: Comparison: Early Literacy Promotion vs Standard Literacy Promotion; Total read scale score between infants at 6 months and 24 months of age in the early literacy arm and the standard literacy arm; Test type: Equivalence — 0.05; p = 0.57, t-test, 2 sided

3. Secondary Outcome: Health Services Utilization
Description: Immunizations and well child visit data will be collected from electronic health records to measure impact of ELP intervention on health services use.
Time Frame: Birth to 6 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | Early Literacy Promotion | Standard Literacy Promotion
Number analyzed (Participants) | 57 | 54
Participants
  Well Child Visits Up to Date | 32 | 40
  Vaccinations Up to Date | 44 | 36
Statistical Analysis 1: Comparison: Early Literacy Promotion vs Standard Literacy Promotion; Number of up to date child well visits between the early literacy arm and the standard literacy arm at 6 months of age; Test type: Equivalence — 0.05; p = 0.23, Chi-squared
Statistical Analysis 2: Comparison: Early Literacy Promotion vs Standard Literacy Promotion; Number of up to date child vaccinations between the early literacy arm and the standard literacy arm at 6 months of age; Test type: Equivalence — 0.05; p = 0.71, Chi-squared

ADVERSE EVENTS:
Time Frame: The All-Cause Mortality Adverse Event for each participant over the 24-month period of participation.
Arm/Group | Early Literacy Promotion | Standard Literacy Promotion
All-Cause Mortality (participants affected / at risk) | 1/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Literacy Promotion (N=60) | Standard Literacy Promotion (N=60)
Mortality (General disorders) | 1 (1) | NA — 1 participant in the ELP arm died of presumed SIDS.

LIMITATIONS AND CAVEATS:
1. Study setting and demographics may not be generalizable to other sites.
2. Participating families in the SLP arm with older children may have been exposed to the ROR program already, likely initiating shared reading prior to 6 months of age.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT02713659/Prot_SAP_000.pdf